CLINICAL TRIAL: NCT01215383
Title: The Antiatherogenic Properties of HDL in Psychiatric Patients With and Without Antipsychotic Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Osamah Hussein, Head of Internal Medicine Department A, Ziv Hospital
Other Study IDs: 0036-10
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: HDL; psychiatric patients; psychiatric patients before and during antipsychotic therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- psychiatric patients: 20 in patients and outpatients with schizophrenia, schizoaffective and bipolar disorder based on psychiatrist diagnostic evaluation using DSM-IV criteria, before and at least two months after antipsychotic therapy will be enrolled.
- healthy volunteers: Ten healthy volunteers will be checked as controls:
  Employee from the hospital staff with no metabolic disease (Diabetes mellitus, hypertension or dyslipidemia) and non-smokers.

SUMMARY:
Background:

Among individuals with schizophrenia, there is an increased prevalence of obesity, dyslipidemia ,diabetes mellitus and related conditions such as cardiovascular disease. People with severe mental illnesses, such as schizophrenia, depression or bipolar disorder, have worse physical health and reduced life expectancy compared to the general population. Number of epidemiological studies of patients with schizophrenia have documented a higher incidence of cardiovascular disease than in the general population, and patients with schizophrenia may be at an elevated risk for cardiovascular disease even in the absence of antipsychotic treatment.

Affinity for the H1 receptor is most closely linked to increased weight gain, although affinity for D2, 5-HT1A, 5-HT2C and a2-receptors may also be involved. Drug affinity for the H1, M3 and 5-HT2C receptors is correlated with an increased risk of diabetes.

High-density lipoprotein cholesterol (HDL-C) concentration in the blood is independently and inversely associated with an increased risk of cardiovascular disease(CVD). However many patients with 'normal' or even 'elevated' plasma HDL experience clinical events. HDL may not always be atheroprotective and in some conditions, it paradoxically enhances the process of atherosclerosis. In addition to its role in reverse cholesterol transport, HDL shows many other protective properties towards atherosclerosis. HDL inhibits the chemotaxis of monocytes , prevents endothelial dysfunction and apoptosis, prohibit slow-density lipoprotein (LDL ) oxidation, and stimulates the proliferation of endothelial cells and smooth muscle cells. These anti-inﬂammatory, antioxidative, antiaggregatory, anti-coagulant, and pro-ﬁbrinolytic activities are exerted by different components of HDL

Aim of the study:

To investigate the functional properties of HDL in psychiatric patients before and during antipsychotic therapy.

Patients and methods:

The blood will be drawn at baseline before the initiation of antipsychotic drugs and 2 months under the antipsychotic treatment.

Study procedures:

Full lipid profile including triglycerides, LDL-C, Total cholesterol, HDL-cholesterol, apo AI, apoAII and apoB100.

Serum Paraoxanase Activity

LDL oxidation and resistance to oxidation (measured by conjugated diens formation during incubation in the presence of copper).

HDL composition: total and unesterified cholesterol, triglycerides and phospholipids, TBARS content before and after exposure to AAPH as a major indicator of oxidative stress, PON activity using phenylacetate as a substrate, apoA1and PAF.

Serum parameters e.g. Diacyl glycerol acyltransferase activity, free ApoA1 and LCAT activity.

3 [H]-Cholesterol efflux will be measured by incubating J744 macrophages with serum. Radioactivity will measured by β counter in the cell lysate and the medium.

Statistical methods:

One-way AVOVA and Student's t-test for paired samples will be used for comparison of multiple groups and paired samples, respectively. p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* in patients and outpatients with schizophrenia, schizoaffective and bipolar disorder based on psychiatrist diagnostic evaluation using DSM-IV criteria, before and at least two months after antipsychotic therapy will be enrolled.

Exclusion Criteria:

* Unwillingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: psychiatric patients before and during antipsychotic therapy
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center (Government Hospital), Safed, Israel